CLINICAL TRIAL: NCT04136327
Title: A Phase 1, Open-label, Single-center Study to Investigate the Pharmacokinetics and Metabolism of GLPG1972 in Healthy Male Subjects Following Single Intravenous [14C]-GLPG1972 Microtracer and Single Oral [14C]-GLPG1972 Administration
Brief Title: A Study in Healthy Male Volunteers to Test How the Test Medicine GLPG1972 is Taken up by the Body When Given by Mouth and Into the Vein as an Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG1972-CL-108; 2019-001305-25 (EudraCT Number)
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLPG1972 oral and [14C]-GLPG1972 IV (Experimental): GLPG1972 film-coated tablet followed by [14C]-GLPG1972 solution for infusion
  Interventions: Drug: GLPG1972 film-coated tablets; Drug: [14C]-GLPG1972 solution for infusion
- [14C]-GLPG1972 oral solution (Experimental): [14C]-GLPG1972 oral solution
  Interventions: Drug: [14C]-GLPG1972 oral solution

INTERVENTIONS:
Drug: GLPG1972 film-coated tablets — single oral dose of GLPG1972
  Arms: GLPG1972 oral and [14C]-GLPG1972 IV
Drug: [14C]-GLPG1972 solution for infusion — a 15-minute IV infusion [14C]-GLPG1972
  Arms: GLPG1972 oral and [14C]-GLPG1972 IV
Drug: [14C]-GLPG1972 oral solution — single oral dose of [14C]-GLPG1972
  Arms: [14C]-GLPG1972 oral solution

SUMMARY:
The sponsor wants to investigate in this study how well the test medicine is taken up by the body when given orally (by mouth) as a tablet and solution, and as a solution for infusion (into a vein). The oral solution and solution for infusion will be radiolabelled. 'Radiolabelled' means that the test medicine has a radioactive component which helps us to track where the test medicine is in the body, what it is broken down into, and how it leaves the body.

The sponsor will also look at the safety and tolerability of the test medicine.

ELIGIBILITY:
Inclusion Criteria:

* Male between 30-64 years of age (extremes included), on the date of signing the Informed Consent Form (ICF).
* A body mass index (BMI) between 18.0-32.0 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and fasting clinical laboratory safety tests. Clinical laboratory safety test results must be within the reference ranges or considered not clinically significant in the opinion of the investigator.
* Having a regular daily defecation pattern (i.e. 1 to 3 times per day).

Exclusion Criteria:

* Known hypersensitivity to IMP ingredients or history of a significant allergic reaction to IMP ingredients as determined by the investigator, and/or known sensitivity to IMP or the excipients (e.g. lactose). Hayfever is allowed unless active.
* History of or a current immunosuppressive condition (e.g. human immunodeficiency virus [HIV] infection).
* Having any illness, judged by the investigator as clinically significant, in the 3 months prior to first investigational medicinal product (IMP) administration.
* Participation in a study with 14C-radiolabeled drug in the last 12 months prior to first IMP administration.
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 millisievert (mSv) in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, can participate in the study.

Ages: 30 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Change of total radioactivity excreted in urine and feces combined (Period 2) | From Day 1 pre-dose up to Day 10
  To assess the mass balance, using [14C]-GLPG1972
Maximum observed plasma concentration (Cmax) of total radioactivity (Period 2) | From Day 1 pre-dose up to Day 10
  To assess the pharmacokinetics (PK) of GLPG1972 and its main metabolites in plasma
Cmax of GLPG1972 (Period 2) | From Day 1 pre-dose up to Day 10
  To assess the PK of GLPG1972 and its main metabolites in plasma
Area under the plasma concentration-time curve (AUC) of total radioactivity (Period 2) | From Day 1 pre-dose up to Day 10
  To assess the PK of GLPG1972 and its main metabolites in plasma
AUC of GLPG1972 (Period 2) | From Day 1 pre-dose up to Day 10
  To assess the PK of GLPG1972 and its main metabolites in plasma
Change in amount of [14C]-GLPG1972 excreted in urine and feces combined (μg) from baseline at Day 7 (Part 2) | From Day 1 pre-dose up to Day 7
  To characterize the elimination pathways and metabolite profile of GLPG1972

SECONDARY OUTCOMES:
Intravenous (IV) Cmax of [14C]-GLPG1972 microtracer (MT)(Period 1) | From Day 1 pre-dose up to Day 4
  To assess the PK of GLPG1972 and its main metabolites in plasma
IV Cmax of total radioactivity (Period 1) | From Day 1 pre-dose up to Day 4
  To assess the PK of GLPG1972 and its main metabolites in plasma
IV AUC of [14C]-GLPG1972 MT (Period 1) | From Day 1 pre-dose up to Day 4
  To assess the PK of GLPG1972 and its main metabolites in plasma
IV AUC of total radioactivity (Period 1) | From Day 1 pre-dose up to Day 4
  To assess the PK of GLPG1972 and its main metabolites in plasma
The number of incidents of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs) and TEAEs leading to discontinuations (Period 1 and Period 2) | From Day 1 through study completion, an average of 2 months
  To evaluate the safety and tolerability of GLPG1972 (Period 1 and Period 2)

CONTACTS AND LOCATIONS:
Overall Officials: Angela de Haas-Amatsaleh, MD, Study Director — Galapagos NV
Locations (1):
- Quotient Sciences Limited, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No